CLINICAL TRIAL: NCT04317417
Title: Using MOST to EMPOWER: Optimizing an Emotion Regulation Intervention to Enhance Well-being Among Adolescents and Young Adult Cancer Survivors
Brief Title: MOST EMPOWER: Optimizing An Emotion Regulation Intervention
Acronym: MOST EMPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00057993; WFBCCC 04220 (Other: Wake Forest Baptist Comprehensive Cancer Center); R01CA242849-01 (NIH)
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Adolescents; Young Adults; Post-treatment cancer survivors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Condition 1 (Experimental): 1) Cognitive Changes after Cancer, 2) Diet, 3) Weight Management, 4) Financial Literacy and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 2 (Experimental): 1) Cognitive Changes after Cancer, 2) Diet, 3) Weight Management, 4) Financial Literacy and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 3 (Experimental): 1) Cognitive Changes after Cancer, 2) Diet, 3) Weight Management, 4) Strengths/ Achievable Goals and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 4 (Experimental): 1) Cognitive Changes after Cancer, 2) Diet, 3) Weight Management, 4) Strengths/ Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 5 (Experimental): 1) Cognitive Changes after Cancer, 2) Diet, 3) Positive Reappraisal , 4) Financial Literacy and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 6 (Experimental): 1) Cognitive Changes after Cancer, 2) Diet, 3) Positive Reappraisal , 4) Financial Literacy and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 7 (Experimental): 1) Cognitive Changes after Cancer, 2) Diet, 3) Positive Reappraisal , 4) Strengths/ Achievable Goals and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 8 (Experimental): 1) Cognitive Changes after Cancer, 2) Diet, 3) Positive Reappraisal , 4) Strengths/ Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 9 (Experimental): 1) Cognitive Changes after Cancer, 2) Mindfulness, 3) Weight Management, 4) Financial Literacy and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 10 (Experimental): 1) Cognitive Changes after Cancer, 2) Mindfulness, 3) Weight Management, 4) Financial Literacy and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 11 (Experimental): 1) Cognitive Changes after Cancer, 2) Mindfulness, 3) Weight Management, 4) Strengths/ Achievable Goals and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 12 (Experimental): 1) Cognitive Changes after Cancer, 2) Mindfulness, 3) Weight Management, 4) Strengths/ Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 13 (Experimental): 1) Cognitive Changes after Cancer, 2) Mindfulness, 3) Positive Reappraisal , 4) Financial Literacy and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 14 (Experimental): 1) Cognitive Changes after Cancer, 2) Mindfulness, 3) Positive Reappraisal , 4) Financial Literacy and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 15 (Experimental): 1) Cognitive Changes after Cancer, 2) Mindfulness, 3) Positive Reappraisal , 4) Strengths/ Achievable Goals and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 16 (Experimental): 1) Cognitive Changes after Cancer, 2) Mindfulness, 3) Positive Reappraisal , 4) Strengths/ Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 17 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Weight Management, 4) Financial Literacy and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 18 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Weight Management, 4) Financial Literacy and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 19 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Weight Management, 4) Strengths/ Achievable Goals and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 20 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Weight Management, 4) Strengths/ Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 21 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Positive Reappraisal , 4) Financial Literacy and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 22 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Positive Reappraisal , 4) Financial Literacy and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 23 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Positive Reappraisal , 4) Financial Literacy and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 24 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Positive Reappraisal , 4) Strengths/ Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 25 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Diet, 3) Positive Reappraisal , 4) Strengths/ Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 26 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Mindfulness, 3) Weight Management, 4) Financial Literacy and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 27 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Mindfulness, 3) Weight Management, 4) Strengths/ Achievable Goals and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 28 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Mindfulness, 3) Weight Management, 4) Strengths/Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 29 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Mindfulness, 3) Positive Reappraisal , 4) Financial Literacy and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 30 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Mindfulness, 3) Positive Reappraisal , 4) Financial Literacy and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER
- Condition 31 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Mindfulness, 3) Positive Reappraisal , 4) Strengths/ Achievable Goals and 5) Sun Protection
  Interventions: Behavioral: EMPOWER
- Condition 32 (Experimental): 1) Positive Events, Capitalizing and Gratitude, 2) Mindfulness, 3) Positive Reappraisal , 4) Strengths/ Achievable Goals and 5) Acts of Kindness
  Interventions: Behavioral: EMPOWER

INTERVENTIONS:
Behavioral: EMPOWER — Participants will receive weekly material for a total of 5 weeks consisting of 1-2 days of didactic content and several days of brief, real-life skills practice and reporting taking approximately 10-15 minutes to complete. Adolescents and young adults cannot skip ahead, but they can return to old lessons or exercises if they choose. Most exercises are done in a "diary" format in which past responses are displayed next to their new ones, so that every time they visit that exercise they see their growing list of past positive experiences. Participants will be permitted up to 8 weeks to complete this self-guided intervention.

SUMMARY:
This purpose of this study is to test a digital health intervention that may promote well-being among young adult cancer survivors. Investigators hope to learn more about wellness and health-related quality of life among young adult cancer survivors by promoting well-being and teaching skills for healthy coping and mood management.

DETAILED DESCRIPTION:
The EMPOWER Intervention is composed of five components:

1. Noting daily positive event, capitalizing on and savoring positive events, and gratitude.
2. Mindfulness
3. Positive Reappraisal
4. Focusing on personal strengths, setting and working toward attainable goals
5. Small of Kindness

For subjects who do not receive EMPOWER components or only receive some of the EMPOWER components, they will be given inert content. The inert content will cover Cognitive changes during Cancer, Diet, Weight Management, Financial Literacy and Sun Protection. The trial is a composed of a full factorial design with 32 (2X2X2X2X2) experimental conditions. Adolescents and Young Adults will receive 0, 1,2,3,4 or 5 Empower components.

Primary Objective

• Identify which of five components in the EMPOWER web based curriculum, contribute meaningfully to positive affect among post-treatment adolescent and young adult cancer survivors.

Secondary Objective

* Identify which of five components in the EMPOWER web based curriculum, contribute meaningfully to depression and anxiety among post-treatment adolescent and young adult cancer survivors.
* Identify which of five components in the EMPOWER web based curriculum, contribute meaningfully to life satisfaction and general self-efficacy among post-treatment adolescent and young adult cancer survivors.

Exploratory Objectives

* Summarize adherence and retention by participants over the course of the EMPOWER intervention.
* Identify which of five components in the EMPOWER web based curriculum, contribute meaningfully to physical functioning, fatigue, satisfaction with social roles and responsibilities.
* Identify which of five components in the EMPOWER web based curriculum, contribute meaningfully to health behaviors (diet, exercise, sedentary behavior, alcohol consumption, cigarette smoking).
* Examine the trajectory of change in positive affect, life satisfaction, general self-efficacy, depression, and anxiety among post-treatment adolescent and young adult cancer survivors post intervention by intervention component.
* Examine coping self-efficacy as a mediator of the relationship between EMPOWER intervention components and positive affect, life satisfaction, depression, and anxiety.
* Examine potential moderators (age, gender, social support, general self-efficacy, stressors, and positive events) of the relationship between EMPOWER intervention components and positive affect, life satisfaction, depression, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand English
* Past history of a cancer diagnosis (excluding basal cell skin carcinoma)
* 15 to 39 years of age at diagnosis of first cancer and currently between the ages of 15 to 39
* Within 0-5 year's post-active treatment for initial diagnosis or recurrence (Note: Maintenance therapy for hematologic or hormonal therapy for breast cancers are not considered "active treatments" for purposes of this study).
* Internet access through a home computer, tablet or smartphone.

Exclusion Criteria:

* Ever been hospitalized for a psychiatric illness
* Currently receiving palliative or hospice care

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 352 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Positive Affect Computer Adaptive Test (CAT) Questionnaire | Baseline up to 4 months after intervention
  Participants will complete a self-reported questionnaire on psychological well being for feelings that reflect a level of pleasurable engagement with the environment, such as happiness, joy, excitement, enthusiasm, and contentment over the past seven days. A mixed model adjusted for baseline to model the value of the outcome (positive affect) at each time point following the intervention. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. There is no fixed minimum or maximum score.
  Average score (50): Represents the national average for the general population. Higher scores (>50): Indicate higher positive affect than the general population. For example, a T-score of 60 is one standard deviation better than the national average.
  Lower scores (<50): Indicate lower positive affect than the general population. A T-score of 40 is one standard deviation worse than the national average.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Questionnaire | Baseline up to 4 months after intervention
  Participants will complete a self-reported questionnaire to capture the negative aspects of anxiety in the past seven days. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. A higher T-score indicates more of the concept being measured, so higher scores correlate with greater anxiety.
  Below 50: Lower than the average anxiety level of the general population. 50: The average anxiety level for the general population.
  Above 50: Higher than the average anxiety level of the general population. The severity can be categorized as follows:
  Less than or equal to 55: Within normal limits. 55-60: Mild anxiety. 60-70: Moderate anxiety. A score of 60 is one standard deviation above the mean.
  > 70: Severe anxiety.
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Questionnaire | Baseline up to 4 months after intervention
  Participants will complete a self-reported questionnaire to capture the negative aspects of depression over the past seven days. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate a greater severity of depressive symptoms.
  T-score of 50: This score indicates no to slight symptoms. T-score of 60: This score indicates at least moderate depression symptoms. T-scores below 50: These scores indicate fewer depressive symptoms than the average person.
  T-scores above 50: These scores indicate more depressive symptoms than the average person.
Patient-Reported Outcomes Measurement Information System (PROMIS) Life Satisfaction Questionnaire | Baseline up to 4 months after intervention
  Participants will complete a self-reported questionnaire to capture the positive (life satisfaction) aspects of emotional health. Raw scores will be converted to T-scores with a mean of 50 and a standard deviation of 10. There is no set minimum or maximum score, scores usually fall within the 20 to 80 range.
  A T-score of 50 indicates a level of life satisfaction that is average for the U.S. general population.
  Higher scores represent higher levels of life satisfaction. Lower scores represent lower levels of life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: John M Salsman, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT04317417/ICF_000.pdf